CLINICAL TRIAL: NCT01740115
Title: Addressing Alcohol/HIV Consequences in Substance Dependence - Boston ARCH Cohort
Brief Title: Boston Alcohol Research Collaboration on HIV/AIDS (ARCH) Cohort
Status: Completed | Type: Observational
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Richard Saitz, Chair, Department of Community Health Sciences, Professor of Community Health Sciences and Medicine, Boston University Schools of Medicine and Public Health, Boston Medical Center
Other Study IDs: U01AA020784 (NIH); U01AA020784 (NIH)
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: HIV Infection; Alcohol Use; Bone Disease; Substance-Related Disorders
Keywords: HIV; Alcohol Use; Bone Disease; Bone Mineral Density; Bone Microarchitecture; Substance Dependence
MeSH Terms: conditions — HIV Infections; Alcohol Drinking; Bone Diseases; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We are storing serum and plasma for future use. We are also storing dried blood spots.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to expand and continue a cohort of HIV-infected adults to establish the longitudinal Boston ARCH Cohort of 250 HIV-infected men and women with current substance dependence or ever injection drug use that have a spectrum of alcohol use; and to determine the effect of alcohol consumption on changes in bone health prospectively in the Cohort.

DETAILED DESCRIPTION:
Unhealthy alcohol use (i.e. the spectrum ranging from heavy drinking that risks health consequences to dependence) is common among HIV-infected persons and is associated with worse health outcomes among people with HIV infection. However, much remains unknown about alcohol-related health effects in those affected by multiple drugs (particularly opioids), or about specific health effects such as detriment to bone. Alcohol use can disrupt bone remodeling by suppressing formation and increasing resorption; heavy alcohol use is associated with both osteopenia (low bone mineral density [BMD]) and incidence of fractures. Osteopenia is common among HIV-infected patients, and fractures are more common in these patients than among adults without HIV infection. Duration of HIV infection has been found to be associated with low BMD, and antiretroviral therapy (ART) also appears to be associated with BMD decline. While bone health is likely affected by HIV infection, ART, alcohol and other drug (e.g. opioid) use (in addition to other known risk factors), the alcohol-osteopenia association among those with HIV infection is not well-characterized. It is not known whether there is an association, the magnitude and nature of that association, and how the relationship is affected by other commonly co-occurring factors (e.g. opioid use, ART).

Accordingly, as part of the Uganda Russia Boston Alcohol Network for Alcohol Research Collaboration on HIV/AIDS (URBAN ARCH) Consortium, we seek to expand and continue a cohort of HIV-infected adults to establish the Boston ARCH Cohort of 250 HIV-infected adults affected by multiple substances and that have a spectrum of alcohol use. This observational prospective cohort study will involve in-person assessments that will take place at 6-month intervals; participants will be followed for a minimum of 1 year and a maximum of 3.5 years. All assessments will include a researcher-administered questionnaire and breath alcohol test. In addition, the baseline assessment and each annual assessment (12, 24 or 36 months after enrollment) will also include: a urine pregnancy test (females only), blood collection, measurement of bone mineral density of the hip and spine (using Hologic QDR 4500W enhanced-array, whole-body, dual-energy radiographic absorptiometry [Bone Densitometer]), and measurement of bone microarchitecture of the wrist and ankle (using Xtreme CT [a device that measures high-resolution three-dimensional peripheral quantitative computed tomography]). We will conduct laboratory tests on blood samples collected at these time points, including tests for 25(OH) vitamin D3 and phosphatidylethanol (PEth). Remaining plasma and serum samples will be stored for future study of bone markers such as: parathyroid hormone, testosterone, carboxy-terminal collagen crosslinks (CTX) (a marker of osteoclast activity), and osteocalcin (osteoblast activity).

In summation, this study will measure the effect of alcohol consumption on changes in bone health prospectively in HIV-infected adults with current substance dependence or ever injection drug use. To our knowledge, no other prospective HIV/bone study has studied these relevant factors simultaneously or used HR-pQCT to assess bone microarchitecture. Data on alcohol risks to bone health is important information for defining risky drinking amounts for people with HIV infection (and for advising such patients accordingly).

ELIGIBILITY:
Inclusion Criteria:

1. Documented HIV antibody by ELISA confirmed by Western Blot or current HIV viral load greater than 10,000 (in any medical record); or HIV antibody by 4th generation ELISA confirmed by a "Multi-Spot" rapid test for discrimination of HIV-1 from HIV-2 infection and, if necessary in the case of discordant results, nucleic acid testing (NAT) for HIV-1; or any other confirmatory pathway approved by the Massachusetts Department of Public Health, U.S. Centers for Disease Control and Prevention, or Boston Medical Center, Center for Infectious Diseases.
2. Current (12-month) substance dependence, determined by using the Mini International Neuropsychiatric Interview (MINI) or ever injection drug use (IDU)
3. Ability to speak English (fluency)
4. At least one contact person who is likely to know whereabouts (to assist with follow-up)

Exclusion Criteria:

1. Under age 18
2. Pregnancy (confirmed by urine test)
3. Plans to leave Boston area in <1 year
4. Inability to consent or understand interview (determined by trained research assistant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects from an existing cohort of HIV-infected adults (Facilitated Access to Substance Abuse Treatment With Prevention and Treatment of HIV [FAST PATH]) who have indicated interest in future studies and patients from HIV clinical care sites will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2012-11; Primary Completion 2016-03 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Annual mean percent change in hip (femoral neck) bone mineral density (g/cm2) | Between study entry and final visit (minimum of 12 months)
  Bone mineral density will be measured using Hologic QDR 4500W enhanced-array, whole-body, dual-energy radiographic absorptiometry scanner and software, version 13.4.2 (Bone Densitometer)

SECONDARY OUTCOMES:
Annual mean percent change in spine (trabecular bone) bone mineral density (g/cm2) | Between study entry and final visit (minimum of 12 months)
  Bone mineral density will be measured using Hologic QDR 4500W enhanced-array, whole-body, dual-energy radiographic absorptiometry scanner and software, version 13.4.2 (Bone Densitometer) Safety Issue?: No
Proportion with bone mineral density decrease of >6% | Between study entry and final visit (minimum of 12 months)
  Bone mineral density will be measured using Hologic QDR 4500W enhanced-array, whole-body, dual-energy radiographic absorptiometry scanner and software, version 13.4.2 (Bone Densitometer)
Proportion with osteopenia (bone mineral density t score -1 to -2.5 SDs compared to a young adult reference population mean) | Between study entry and final visit (minimum of 12 months)
  Bone mineral density will be measured using Hologic QDR 4500W enhanced-array, whole-body, dual-energy radiographic absorptiometry scanner and software, version 13.4.2 (Bone Densitometer)
Proportion of osteoporosis (bone mineral density t score <-2.5 SDs compared to a young adult reference population mean) | Between study entry and final visit (minimum of 12 months)
  Bone mineral density will be measured using Hologic QDR 4500W enhanced-array, whole-body, dual-energy radiographic absorptiometry scanner and software, version 13.4.2 (Bone Densitometer)
Fractures (vertebral, hip, wrist) | 12 months prior to study entry through final visit
  Self-report of ever fracture at each site (vertebral, hip, wrist) and fracture in past 12-months collected at baseline and each annual time point.
Annual mean percent change in bone mineral density (g/cm2) at site with lowest bone mineral density (spine [trabecular bone] or hip [femoral neck]) | Between study entry and final visit (minimum of 12 months)
  Bone mineral density will be measured using Hologic QDR 4500W enhanced-array, whole-body, dual-energy radiographic absorptiometry scanner and software, version 13.4.2 (Bone Densitometer)

OTHER OUTCOMES:
Bone mineral density, bone mineral content, trabecular thickness, separation and number, volume fraction and cortical thickness | Between study entry and final visit (minimum of 12 months)
  Exploratory outcomes will be assessed using HR-pQCT (wrist and ankle)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Saitz, MD, MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States